CLINICAL TRIAL: NCT01254110
Title: Physiological Study on Glutamine and Leucine Effects on Intestinal Protein Metabolism
Brief Title: Amino Acid and Intestinal Protein Metabolism : Working Study
Acronym: Intesmetapro
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2007/142/HP; ID RCB 2008-A00692-53
Record Dates: First submitted 2009-03-09; First posted 2010-12-06 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Transduction Pathway; Proteinic Synthesis; Proteolytic System

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood duodenal tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Enterally fed with leucine
- 2: Enterally fed with glutamine
- 3: Enterally fed with protein powder

SUMMARY:
Gut protein metabolism that could be influenced by protein supply is involved in the regulation of several physiological functions such as gut barrier function and represents a major contribution in the whole-body protein turnover. Intracellular pathways implicated in the transduction of amino acids effects remained unknown in the human gut. Thus, the aim of the present project is to evaluate and to understand the effects of amino acids (glutamine, leucine) on gut protein metabolism (synthesis and degradation) in young healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* volunteers with seronegativity for HIV1 and HIV2 and HCV and HVB
* good nutritional state with physical indication mass included between 18,5 and 25kg/m2
* non-smoking volunteers
* volunteers without digestive, allergic or haemorrhagic history
* volunteers without progressive disease
* digestive endoscopy tolerance
* age >=18 and <= 50years
* consent obtained from volunteers

Exclusion Criteria:

* smoking volunteers
* volunteers with digestive, or allergic history
* volunteers with haemorrhagic sign
* pregnancy
* progressive digestive disease
* significant progressive disease
* volunteers with therapeutic treatment (aspirin)
* digestive endoscopy intolerance
* volunteers with neurological disorder or with delicate psychological state

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
assessment of intestinal protein synthesis stimulation by Leucine or glutamine in duodenal biopsy | 18 months

SECONDARY OUTCOMES:
Assessment of involved signaling pathways | 18 months
Assessment of intestinal proteolysis | 18 months
Assessment of protein synthesis rate in intestinal mitochondria | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Moise COEFFIER, Study Chair — UH Rouen; Anne-Françoise CAILLEUX, Doctor, Study Chair — UH Rouen
Locations (1):
- Centre d'Investigation Clinique - Hôpital charles Nicolle, Rouen, Seine maritime, France

REFERENCES:
- [Derived] Goichon A, Bertrand J, Chan P, Lecleire S, Coquard A, Cailleux AF, Vaudry D, Dechelotte P, Coeffier M. Enteral delivery of proteins enhances the expression of proteins involved in the cytoskeleton and protein biosynthesis in human duodenal mucosa. Am J Clin Nutr. 2015 Aug;102(2):359-67. doi: 10.3945/ajcn.114.104216. Epub 2015 Jun 24. PMID 26109581
- [Derived] Bertrand J, Goichon A, Chan P, Azhar S, Lecleire S, Donnadieu N, Vaudry D, Cailleux AF, Dechelotte P, Coeffier M. Enteral glutamine infusion modulates ubiquitination of heat shock proteins, Grp-75 and Apg-2, in the human duodenal mucosa. Amino Acids. 2014 Apr;46(4):1059-67. doi: 10.1007/s00726-014-1670-x. Epub 2014 Jan 22. PMID 24449167
- [Derived] Coeffier M, Claeyssens S, Bole-Feysot C, Guerin C, Maurer B, Lecleire S, Lavoinne A, Donnadieu N, Cailleux AF, Dechelotte P. Enteral delivery of proteins stimulates protein synthesis in human duodenal mucosa in the fed state through a mammalian target of rapamycin-independent pathway. Am J Clin Nutr. 2013 Feb;97(2):286-94. doi: 10.3945/ajcn.112.046946. Epub 2013 Jan 2. PMID 23283505
- [Derived] Coeffier M, Claeyssens S, Bensifi M, Lecleire S, Boukhettala N, Maurer B, Donnadieu N, Lavoinne A, Cailleux AF, Dechelotte P. Influence of leucine on protein metabolism, phosphokinase expression, and cell proliferation in human duodenum1,3. Am J Clin Nutr. 2011 Jun;93(6):1255-62. doi: 10.3945/ajcn.111.013649. Epub 2011 Apr 20. PMID 21508089